CLINICAL TRIAL: NCT04606160
Title: Utilizing A Single Session Problem-Solving Intervention With Caregivers of Pediatric Patients Receiving Chronic Transfusion to Treat Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Medical Center Dallas (Other)
Responsible Party: Principal Investigator, Dennis Burchette, Doctoral Student, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU-2020-0181
Record Dates: First submitted 2020-10-21; First posted 2020-10-28 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; chronic transfusion; problem solving; single session intervention; children; pediatrics; pediatric patients; caregivers; scd; intervention; chronic blood transfusion; hematology; sickle cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Session Problem-Solving Intervention (Experimental): Participants will receive a single session problem-solving intervention during visit 2 of the 4 visit research study. During visit 3, participants will receive a review of the intervention from visit 2. During visits 1, 3, and 4, participants will complete measures.
  Interventions: Behavioral: Single Session Problem-Solving Intervention
- Control - Non Single Session Problem-Solving Intervention (No Intervention): These participants will complete measures at visits 1,2,3, and 4. They will also receive a visit during visit 2 of the 4 visit study, where they will only complete measures.

INTERVENTIONS:
Behavioral: Single Session Problem-Solving Intervention — The intervention will be a researcher led 30-45 minute session using the problem-solving module from the Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Issues (MATCH-ADTC protocol.
  Arms: Single Session Problem-Solving Intervention

SUMMARY:
This study seeks to utilize an innovative approach of a single session problem-solving intervention to address psychosocial factors affecting patient outcomes within the pediatric sickle cell population. The study will be a randomized control trial of a single session problem-solving intervention.

This original research will investigate the feasibility and efficacy of utilizing a single-session problem-solving intervention to address problems affecting children and families receiving chronic blood transfusions for sickle cell disease in order to: 1) contribute to literature related to single session problem solving interventions with the chronic transfusion sickle cell population and 2) identify a model of sustainable care that reduces the burden of a multiple session intervention and increases access to services. Additionally, this research aims to provide relatively low burden and potentially highly effective intervention into regular care for this population in order to evaluate the feasibility of integrating a single-session problem solving intervention into routine clinical flow, thereby addressing needs more systematically that have been identified by families. Further, this research aims to identify potential utility of medical providers being trained on providing the intervention, which could be part of a future study.

DETAILED DESCRIPTION:
In the event that research must be completed virtually due to coronavirus (COVID-19) restrictions at the research site, an Ipad will be provided to participants by clinic staff to complete measures, through Research Electronic Data Capture (REDCap) and the intervention/control visits through a Children's Health-approved and HIPAA compliant telehealth platform. Due to continued changes in protocols, it is possible that participants may begin with in-person research and transition to virtual research, or vice versa.

Patient list for chronic blood transfusion clinic will be reviewed weekly for eligible participants. Eligible participants will be approached at the start of their routine blood transfusion (which are part of their clinical care) appointment to minimize interference from sedative medications. The researcher will explain the study and answer questions related to participation. If the caregiver and youth choose to participate, written consent (and patient assent when appropriate) will be obtained.

At visit one, both study groups will receive a baseline visit (V1), which will include completing measures, and participants will be provided a handout of community mental health resources to have for future reference if mental health needs arise. During visit two (V2), (typically occurs approximately 1 month after V1) caregivers in the intervention group will complete the Psychological Outcomes Profiles (PSYCHLOPS) measure, receive a single session problem-solving intervention to target an identified problem, and complete the Abbreviated Acceptability Rating Profile (AARP) at the end of the intervention. Problem to be targeted will be identified collaboratively by the researcher and the caregiver, after review of measures completed by the caregiver and youth participant during visit one. The control group will receive a visit from the researcher, in which the caregiver participant will complete the PSYCHLOPS measure. During visit three (V3), (typically occurs approximately 2 months after V1), both groups will complete the same measures from visit one, with the addition of all caregiver participants completing the PSYCLOPS measure. At this visit, caregivers in the intervention group will also receive a short review of the problem-solving strategy and address questions about the skill following completion of measures. The caregiver participants in the intervention group will complete the AARP at the end of the intervention review. At visit four (V4), (typically occurs approximately five months after V1) both groups will complete the same measures as visit one, in addition to the PSYCHLOPS measure, for longer-term follow up. In addition, the intervention group will complete the AARP.

Virtual alternative for all visits:

All study procedures will remain the same as stated above, except clinic staff will provide the handout of community mental health resources to participants and visits with both the Intervention Group and Control Group will be conducted through a Children's Health-approved telehealth platform.

Aims and Hypotheses

Aim 1: Determine the feasibility of utilizing a single-session problem solving intervention.

Hypothesis 1: At least 70% of participants approached for this study will agree to enroll.

Hypothesis 2: At least 70% of participants who start the study will be retained through V4.

Aim 2: Determine the acceptability of a single-session problem solving intervention.

Hypothesis 3: At least 70% of caregivers will find the single-session intervention to be acceptable at V3.

Hypothesis 4: At least 70% of caregivers will find the single-session intervention to be acceptable at V4.

Aim 3: Determine the efficacy of a single-session problem solving intervention at improving the selected problem.

Hypothesis 5: The intervention group will report a greater decrease in difficulty associated with their identified problem [Psychosocial Outcomes Profiles (PSYCHLOPS)] over time (V3 and V4) compared to those in the control group.

Hypothesis 6: The intervention group will report a greater decrease in psychosocial risk factor score [Psychosocial Assessment Tool (PAT)] over time as compared to the control group.

Hypothesis 7: The intervention group will report a greater increase in quality of life [Pediatrics Quality of Life_ Sickle Cell Disease Module (PedsQL_SCD Module)], both patient and caregiver report) over time as compared to the control group.

ELIGIBILITY:
Patient and Caregiver Participants:

Inclusion Criteria:

* English speaking
* Patient and/or caregiver of patient between the ages of 7 years to less than 19 at time of enrollment
* Patient and/or caregiver of patient diagnosis of sickle cell disease with sickle cell - SS genotype
* Patient and/or caregiver of patient who has received chronic blood transfusions for at least 6 months and continuing through the duration of the study
* Caregiver and patient pair agree to both participate in the study

Exclusion Criteria:

* Patient or caregiver of patient who are temporarily on blood transfusions for a transient complication (e.g., priapism or recurrent acute chest syndrome)
* Patient and/or caregiver of patient displaying clinically evident cognitive delay (e.g., stroke with severe cognitive deficits, intellectual disability) that would preclude completion of measures or participation in intervention as defined by the medical team, researcher, or psychologist.
* Patient and/or caregiver of patient who is a ward of state

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of utilizing the intervention as measured by the number of participants who are eligible and enroll in the study | Time of enrollment, approx. 2-3 days from initial recruitment attempt
  Feasibility of utilizing the intervention will be measured by counting the number of participants who meet the eligibility criteria and enroll in the study
Feasibility of utilizing the intervention as measured by the number of participants who enrolled and were retained through Visit 4. | Time of enrollment until completion of study, approx. 12 months
  Feasibility of utilizing the intervention as measured by counting the number of participants who enrolled and were retained through Visit 4.

SECONDARY OUTCOMES:
Acceptability of the intervention as measured by the number of participants who find an intervention to be acceptable at visit 3 | Following the intervention to visit 3, approx. 1 month from the intervention
  Acceptability will be measured by the AARP (Abbreviated Acceptability Rating Profile) questionnaire.
  AARP created to be an abbreviated form of the Intervention Rating Profile (Witt & Elliott, 1985). The AARP (Tarnowski & Simonian, 1992) was developed as an eight-item measure that is rated on a 6-point Likert scale ranging from one (strongly disagree) to six (strongly agree). Higher scores represent higher acceptability of the intervention. The AARP has a Cronbach's alpha of .97 (Tarnowski & Simonian, 1992).
Acceptability of the intervention as measured by the number of participants who find an intervention to be acceptable at visit 4 | Following the intervention to visit 4, approx. 4 months from the intervention
  Acceptability will be measured by the AARP (Abbreviated Acceptability Rating Profile) questionnaire.
  AARP created to be an abbreviated form of the Intervention Rating Profile (Witt & Elliott, 1985). The AARP (Tarnowski & Simonian, 1992) was developed as an eight-item measure that is rated on a 6-point Likert scale ranging from one (strongly disagree) to six (strongly agree). Higher scores represent higher acceptability of the intervention. The AARP has a Cronbach's alpha of .97 (Tarnowski & Simonian, 1992).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Burchette, Principal Investigator — Doctoral Student Researcher; Jenna Oppenheim, PsyD, Study Chair — Psychologist; Julie Germann, PhD, Study Chair — Psychologist
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared will be deidentified results of the study, including information about feasibility, acceptability, and efficacy data on use of a single session problem-solving intervention use with caregivers of pediatric patients receiving chronic transfusion to treat sickle cell disease.
Supporting Information: SAP
Time Frame: Data will become available when published in journals to contribute to the literature.